CLINICAL TRIAL: NCT04875585
Title: Phase II Trial Exploring Combined Neoadjuvant Therapy With Pembrolizumab/Lenvatinib and Adjuvant Pembrolizumab in Patients With Surgically Resectable Non-Small- Cell Lung Cancer (NSCLC)
Brief Title: Trial Exploring Combined Neoadjuvant Therapy With Pembrolizumab/Lenvatinib + Adjuvant Pembrolizumab in Pat. With NSCLC
Acronym: INNWOP1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Georg Pall, Principal Investigator, Medical University Innsbruck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNWOP2020
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy; pembrolizumab; lenvatinib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): neoadjuvant therapy with Pembrolizumab/Lenvatinib in combination with surgical resection of primary tumor followed by adjuvant Pembrolizumab therapy
  Interventions: Drug: neoadjuvant therapy with Pembrolizumab/Lenvatinib; Procedure: Surgery; Drug: Adjuvant Treatment Phase

INTERVENTIONS:
Drug: neoadjuvant therapy with Pembrolizumab/Lenvatinib — Neoadjuvant therapy for 6 weeks
Procedure: Surgery — surgical resection of primary tumor and lymph-node-dissection.
Drug: Adjuvant Treatment Phase — Adjuvant treatment with 15 cycles of Pembrolizumab

SUMMARY:
The primary aim of this single arm, phase II study is to determine the efficacy of the combination therapy Pembrolizumab/Lenvatinib regarding the rate of major pathological response (MPR-Rate). The investigators expect to improve the MPR-Rate of 20% in Anti-PD1/-PD-L1 monotherapy (observed in recent trials) to a MPR-Rate of 40% with the combination therapy Pembrolizumab/Lenvatinib.

DETAILED DESCRIPTION:
In Tyrol lung cancer is the fourth most incident cancer in women and the second most in men (1). Mortality related to lung cancer is highest in both sex groups, which supports the huge unmet medical need for improved lung cancer therapies in the near future (2). In very recent years, many novel therapies have entered the clinical scene, particular for treatment of non-small cell lung cancer (NSCLC) and many of those drugs target the tumor microenvironment (TME) (3-6). Both, anti-angiogenic-treatment (AAT) and immunotherapy target the TME and have been successfully established as standard therapeutic options in NSCLC (6-9). Recent preclinical studies strongly suggest that AAT and immune-checkpoint-inhibitors act synergistically and first clinical studies also proved an acceptable safety profile (6, 10, 11).

However, response and therapeutic efficacy of these approaches is still limited to certain subgroups of patients and therefore the search for biomarker(s) predicting response and/or toxicity for improved patient selection is of utmost importance. This knowledge would definitely allow a more rational and efficient clinical use of these compounds. Neoadjuvant "window of opportunity" trials may offer an important way of answering relevant translational research questions related to optimized (biomarker-driven) patient selection, as they allow sequential tissue sampling during diagnostic work-up and subsequently (after neoadjuvant therapy) upon surgical tumor resection. Most studies investigating immunotherapy combinational approaches mainly focused on the characterization of the immune cell compartment, while the influence on the vascular network as well as on their mutual regulation, particularly in case both compartments are targeted in parallel, has not sufficiently been addressed.

Standard neoadjuvant therapy is a mainstay of combinational chemotherapy with high toxicity and complication rates (12, 13). Several recent early clinical trials have shown promising pathologic response rates and good tolerability with neoadjuvant immune-checkpoint antibody therapy (14-16). Recently, neoadjuvant immune-checkpoint antibody monotherapy (ICA) with the PD-1 blocking monoclonal antibody Nivolumab showed high pathological response rates and good tolerability (14).

Adjuvant treatment with immune-checkpoint-inhibitors has been shown to be effective and safe in the treatment of early stage melanoma (17, 18). In NSCLC prospective randomized trials with the aim of recapitulating these beneficial effects are ongoing. A high medical need in the adjuvant therapy setting is to select the optimal candidates for therapy and liquid-biopsies drawn during adjuvant treatment offer important opportunities for patients selection: (i) the kinetics of cell-free tumor-DNA (ct-DNA) can be used to monitor remission status and potentially early sense later overt clinical relapse (19-22); (ii) longitudinal assessment of patient-specific tumor alterations may predict therapy recurrence (iii) together with measurements of immune cell populations ct-DNA kinetics might gain insights into the dynamics within the TME during a prolonged period of checkpoint-blockade. Combining these informations might lead to a better understanding of potentially beneficial neo-/adjuvant treatment effects finally leading to relapse-prevention.

The present phase II investigator-initiated trial (IIT) investigates the efficacy of the neoadjuvant combination therapy of the PD-1 inhibitor Pembrolizumab with the antiangiogenic kinase inhibitor Lenvatinib (primary endpoint: major pathological response) and how this therapy shapes the TME. Furthermore, the disease kinetics and the effects on cellular and soluble immune-biomarkers will be monitored during an additional adjuvant treatment-phase with Pembrolizumab via liquid-biopsies, multi-dimensional flow cytometry and cytokine quantification. In total 33 patients with early stage NSCLC will be included in this trial. The scientific program provides a comprehensive mapping of the TME prior to and after neoadjuvant intervention using various single cell analysis platforms to depict the composition of the TME. Consecutively collected plasma and blood probes will be analysed and correlated with routine response assessment, TME patterns and the clinical endpoints.

In conclusion, the present phase II study aims for identification of potential biomarkers and biomarker combinations relevant for combination therapy of immunotherapy and anti-angiogenic agents in early stage NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants ≥18 years of age
2. Histologically confirmed primary diagnosis of resectable NSCLC, stages IA3-IIIA (max. single station N2).
3. Measurable disease based on RECIST 1.1.
4. Male participants must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 additional days after the last dose of study treatment and refrain from donating sperm during this period.
5. Female participants are eligible to participate if not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
6. Written informed consent provided
7. ECOG performance status of 0 to 1
8. Adequate organ function. Specimens must be collected within 14 days prior to the start of study treatment.

Exclusion Criteria:

1. A woman with child-bearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to inclusion (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Uncontrolled blood pressure (systolic BP>160mmHg or diastolic BP >95mmHg) despite an optimized regimen of antihypertensive medication.
3. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, and/or cardiac arrhythmia requiring medical treatment at screening.
4. History of prolonged QT syndrome, or family member with prolonged QT syndrome
5. QTc interval >490 msec when 3 consecutive ECG values are averaged
6. Bleeding and/or thrombotic disorders and/or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following Lenvatinib therapy.
7. Subjects having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
8. Patient has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (eg, CTLA-4, OX 40, CD137).
9. Patient has received prior systemic anti-cancer therapy for the newly diagnosed NSCLC including investigational agents.
10. Patient has received prior radiotherapy for the newly diagnosed NSCLC.
11. Patient has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
12. Patient is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
13. Diagnosis of immunodeficiency and/or patient is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
14. Known additional malignancy that is progressing.
15. Known history of severe (≥Grade 3) allergic or hypersensitivity reactions to Pembrolizumab or Lenvatinib and/or any of their excipients.
16. Known active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
17. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
18. Active infection requiring systemic therapy.
19. Infection with Human Immunodeficiency Virus (HIV).
20. Infection with Hepatitis B and/or Hepatitis C
21. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Patient has received prior surgery therapy for the newly diagnosed NSCLC.
23. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Major pathological response after neoadjuvant immunotherapy in combination with angiogenesis inhibition | 2 years
  Number of Participants Reaching a Major Pathological Response after Short Course Neoadjuvant Treatment with Pembrolizumab/Lenvatinib.

SECONDARY OUTCOMES:
Radiologic response according to RECIST/iRECIST | 2 years
Surgical resection rate | 2 years
Disease free survival at 1, 2, 3 and 5 years | 5 years
Overall survival at 1, 2, 3 and 5 years | 5 years
Capturing of the Toxicity of a neoadjuvant/adjuvant treatment | 5 years
  Capturing of the Toxicity of a Neoadjuvant Treatment with Pembrolizumab/Lenvatinib and Adjuvant Pembrolizumab (Common Toxicity Criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Georg Pall, Dr., Principal Investigator — Georg.Pall@i-med.ac.at
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No